CLINICAL TRIAL: NCT04710693
Title: Implementation of Optical Diagnosis of Diminutive Colorectal Polyps in Real Life Clinical Practice: DISCARD3 Study (Incorporating AI-DETECT)
Brief Title: Implementation of Optical Diagnosis of Diminutive Colorectal Polyps: DISCARD3 Study (Incorporating AI-DETECT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 245862
Record Dates: First submitted 2020-12-14; First posted 2021-01-15 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-09

CONDITIONS: Colonic Polyp
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Intervention Model Description: Colonoscopy lists will be randomised for the use of a CAD polyp-detection system to be used as an adjunct to optical diagnosis. 50% of colonoscopy lists will be randomly assigned to use the CAD system and 50% of colonoscopy lists will not use the CAD system.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAD polyp-detection system (Other): In this arm, a CAD polyp detection system will be used during the colonoscopy.
  Interventions: Diagnostic Test: CAD polyp-detection system
- Standard (no CAD polyp-detection system) (No Intervention): In this arm, a CAD polyp detection system will not be used during the colonoscopy.

INTERVENTIONS:
Diagnostic Test: CAD polyp-detection system — Software will be used during the procedure to aid the detection of polyps during the procedure.
  Arms: CAD polyp-detection system

SUMMARY:
This is a prospective feasibility study. The aim of this work is to assess the acceptability and feasibility of optical diagnosis-led care in bowel cancer screening patients undergoing colonoscopy. This study will determine whether bowel cancer screening colonoscopists are able to consistently record and diagnose diminutive adenomas suitable for a resect and discard strategy allowing assignment of surveillance intervals according to Preservation and Incorporation of Valuable Endoscopic Innovations (PIVI) criteria. A practical quality assurance program around optical diagnosis will be introduced. The use of a CAD polyp-detection system will also be evaluated (AI-DETECT).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 60-74

  * with +ve Faecal Occult Blood/Faecal Immunochemical test attending for screening colonoscopy within BCSP (Bowel Cancer Screening Programme)
  * with an established history of adenomas attending for surveillance colonoscopy within BCSP
* Patients aged 55 - referred for screening colonoscopy following positive Bowel Scope Screening flexible sigmoidoscopy

Exclusion Criteria:

* Patients with a risk profile (due to family history or other) whose follow-up will be outside standard BCSP
* Patients with inflammatory bowel disease
* Unable to consent
* Pregnancy

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Learning curve to achieve accurate optical diagnosis | Through study completion, approximately 18-24 months
  The investigators will assess endoscopist learning curve by calculating percentage of accurate optical diagnoses of diminutive polyps (when compared with histopathology) for all endoscopists over the course of the study.
Proportion of cases where optical diagnosis derived surveillance intervals concur with histopathology derived surveillance intervals | 2 weeks for each participant
  For each participant, the surveillance interval according to international guidelines (UK, US, European) will be determined based on optical diagnoses alone and then separately based on histopathology results alone. The proportion of cases where both optical diagnosis derived and histopathology derived surveillance intervals agree will be calculated.
Polyp detection rate (AI-DETECT) | 2 weeks for each participant
  The investigators will assess the impact on polyp detection rate when using a CAD polyp-detection system.

SECONDARY OUTCOMES:
Sensitivity of optical diagnosis | 2 weeks for each participant
  The sensitivity of optical diagnosis will be assessed for polyps identified during the course of the study.
Specificity of optical diagnosis | 2 weeks for each participant
  The specificity of optical diagnosis will be assessed for polyps identified during the course of the study.
Adenoma detection rate (AI-DETECT) | 2 weeks for each participant
  The investigators will assess the impact on adenoma detection rate when using a CAD polyp-detection system.
Serrated polyp detection rate (AI-DETECT) | 2 weeks for each participant
  The investigators will assess the impact on serrated polyp detection rate when using a CAD polyp-detection system.

CONTACTS AND LOCATIONS:
Locations (1):
- St Mark's Hospital, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahmad A, Moorghen M, Wilson A, Stasinos I, Haycock A, Humphries A, Monahan K, Suzuki N, Thomas-Gibson S, Vance M, Thiruvilangam K, Dhillon A, Saunders BP. Implementation of optical diagnosis with a "resect and discard" strategy in clinical practice: DISCARD3 study. Gastrointest Endosc. 2022 Dec;96(6):1021-1032.e2. doi: 10.1016/j.gie.2022.06.019. Epub 2022 Jun 18. PMID 35724693